CLINICAL TRIAL: NCT06899425
Title: Effect of Kinesio Tape on Neck Pain in Lactating Women. A Randomized Controlled Trial
Brief Title: Effect of Kinesio Tape on Neck Pain in Lactating Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Asem Abd El-Ghaffar Amr, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003812
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain Musculoskeletal
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot pack group (Active Comparator): The participants will be treated by hot packs on the neck for 12 weeks.
  Interventions: Other: Hot pack
- kinesio tape and hot pack group (Experimental): The participants will be treated by hot packs and kinesio tape on the neck for 12 weeks.
  Interventions: Other: Hot pack; Other: Kinesio tape

INTERVENTIONS:
Other: Hot pack — The participants will be treated by hot packs on neck for 15 minutes, 3 times per weeks for 12 weeks.
Other: Kinesio tape — The participants will be treated by hot packs and kinesio tape. The tape will be placed for several days (3-5 days of application) then it will be removed and repeated for 12 weeks.
  Arms: kinesio tape and hot pack group

SUMMARY:
This study will be conducted to investigate the effect of kinesio tape on neck pain in lactating women.

DETAILED DESCRIPTION:
Neck pain is widely prevalent and can be exacerbated by poor posture and prolonged or repetitive positions-both of which are common in lactating mothers. Research shows that a significant percentage of breastfeeding women experience musculoskeletal pain, often linked to specific postures such as the cross-cradle hold. Prolonged forward head posture (FHP) and muscle imbalances in the neck-shoulder region further contribute to mechanical neck pain by placing excessive strain on muscles, joints, and connective tissues.

Kinesio taping (KT) is a non-pharmacological technique aimed at alleviating pain and improving functional movement. By lifting the skin slightly, KT is proposed to enhance local blood and lymphatic flow, reduce nociceptive signals, and stimulate proprioceptive feedback. Multiple studies suggest KT can help correct posture, relieve muscle fatigue, and improve range of motion, thus offering a promising intervention for mechanical neck pain. These benefits are potentially valuable for lactating mothers, who are especially prone to postural stresses and neck discomfort due to the physical demands of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* All women are complaining from neck pain.
* Their ages will be ranged from 20 to 30 years old.
* Their body mass index will not exceed 30 kg/m².
* They are medically stable and consented to participate in the study.

Exclusion Criteria:

* Cervical spondylosis.
* Cervical disc prolapse.
* History of fracture of cervical spine.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-03-29 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 12 weeks
  Pain will be assessed through visual analogue scale (VAS) for each woman in both groups before and after treatment. It is usually a horizontal line, 100 mm long, whose ends are labeled as the extreme ("no pain" and "pain as bad as it could be"). The patient is asked to put a mark on the line indicating their pain intensity. Sometimes descriptive, such as 'mild', 'moderate', 'sever', or numbers are provided along the scale for guidance. it is valid and reliable tool to assess pain intensity.
Pain pressure threshold | 12 weeks
  An electronic pressure algometer "Force one gauge- model FDI" (Wagner instruments, Greenwish, CT, USA) will be used to measure myofascial trigger points tenderness by determining the pain pressure threshold using a pressure probe, that's placed on the trigger point. With a 1-cm 2 rubber disc at the end of the device. Pressure will be applied perpendicularly to the skin at constant speed, and the woman will be asked to say stop at the time she started feeling pain.

SECONDARY OUTCOMES:
Neck flexion range of motion | 12 weeks
  Goniometer will be used to measure neck flexion range of motion for all women in both groups before and after treatment. The axis of the goniometer will be placed over the external auditory meatus. The stationary arm placed vertically or perpendicular to the floor and the moving arm placed on the base of the nose. The participants will be asked to flex neck and the angle will be recorded. Normal cervical flexion range of motion is usually approximately 80º.
Neck extension range of motion | 12 weeks
  Goniometer will be used to measure neck extension range of motion for all women in both groups before and after treatment. The axis of the goniometer will be placed over the external auditory meatus. The stationary arm placed vertically or perpendicular to the floor and the moving arm placed on the base of the nose. The participants will be asked to extend neck and the angle will be recorded. Normal cervical extension range of motion is usually approximately 50º.
Neck lateral flexion range of motion | 12 weeks
  Goniometer will be used to measure neck extension range of motion for all women in both groups before and after treatment. The axis of the goniometer will be placed over the spinous process of the C7. The stationary arm placed along the imaginary line between the two acromion processes either vertically or perpendicular to the floor or horizontal and parallel to the floor and the moving arm placed over the external occipital protuberance. The participants will be asked to perform lateral flexion of the neck and the angle will be recorded. Normal cervical lateral flexion range of motion is usually approximately 45º.
Neck rotation range of motion | 12 weeks
  Goniometer will be used to measure neck extension range of motion for all women in both groups before and after treatment. The axis of the goniometer will be placed over the over to the center of the patients' head. The stationary arm placed along an imaginary line between the two acromion processes and the moving arm placed at the tip of the nose. the participants will be asked to perform neck rotation and the angle will be recorded. Normal cervical rotation range of motion is usually approximately 80º.
Northwick park neck pain questionnaire | 12 weeks
  A neck pain questionnaire using nine five-part sections has been devised to overcome this problem. Questions on duration and intensity of pain were good indicators of a patient's global assessment. The questionnaire is easy for patients to complete, simple to score and provides an objective measure to evaluate outcome in patients with acute or chronic neck pain. The questionnaire consists of 9 sections about daily activities. Each section contains 1 question and 5 statements. Each section is scored on a 0-4 scale, 4 representing the greatest disability, and 0 representing the least disability. The total score is obtained by summing the scores for the 9 sections (possible score: 0-36).

CONTACTS AND LOCATIONS:
Overall Officials: Abd El Hamid Atta Allah, PHD, Study Director — Al-Azhar University; Mohamed Awad, Professor, Study Chair — Cairo University
Locations (1):
- Al Zahra University Hospital, Cairo, Egypt